CLINICAL TRIAL: NCT05864820
Title: The Use of Photogrammetric Technology for the Evaluation of Anthropometric Measurements and Body Composition
Brief Title: Photogrammetric Scan System for Body Composition Analysis
Status: Terminated | Type: Observational
Why Stopped: Inability to continue corporate collaboration for analysis for body composition analysis through photogrammetric scan system.
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: AVATARGET (PI: M Briguglio); L3052 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Anthropometry; Musculoskeletal System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational study evaluates the goodness of the IGOODI photogrammetric scan system in measuring anthropometry and estimating the body composition of 75 healthy subjects, comparing the results with the measurements taken using methods used in clinical practice, including body circumferences and bioimpedance analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female gender
* Between the ages of 18 and 85
* Caucasian race
* Cognitively intact
* Acceptance and signing of informed consent
* Height between 120 and 200 cm (included)

Exclusion Criteria:

* Congenital or acquired musculoskeletal deformities of the limbs or trunk
* Implants resulting from cosmetic surgery
* Articular prostheses and/or means of synthesis
* Current oncological or metabolic pathologies
* Photosensitivity
* Epilepsy
* Claustrophobia
* Subjects unable to independently maintain an upright position
* Wearers of pacemakers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects of the general population
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Correlation between anthropometric circumferences | Baseline and after 1 year
  Association between the circumferences taken with clinical practice methodology (inelastic and flexible tape measure) and the results from the photogrammetric technology

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Briguglio, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided